CLINICAL TRIAL: NCT03490916
Title: A Prospective, Double-blind, Randomized, Placebo-controlled Trial of Acetazolamide on Subclinical High-Altitude Pulmonary Edema Detected by Lung Ultrasonography
Brief Title: Effect of Acetazolamide on Subclinical High-Altitude Pulmonary Edema Detected by Lung Ultrasonography
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI was unable to continue to gather data during the trip during to medical illness
Sponsor: Vincent Kan (Other)
Responsible Party: Sponsor-Investigator, Vincent Kan, Former Fellow, Department of Emergency Medicine, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H00014860
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: High Altitude Pulmonary Edema
Keywords: Acetazolamide; High-altitude illness; High-altitude pulmonary edema; Lung comets; Lung ultrasound; Subclinical high-altitude pulmonary edema
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetazolamide normal dose (Experimental): One (1) dose of 250mg of Acetazolamide
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): One (1) dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Administration of Acetazolamide
  Other Names: diamox
  Arms: Acetazolamide normal dose
Drug: Placebo — Administration of Placebo
  Arms: Placebo

SUMMARY:
The overall goal of this study is to detect preclinical signs of HAPE by lung ultrasonography and evaluate the effectiveness of acetazolamide at decreasing pulmonary edema by using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Able to consent
3. English speaking
4. Trekking directly to Everest Base Camp

Exclusion Criteria:

1. Age less than 18 years
2. Non-English speaking
3. Pregnant
4. Already had a diagnosis of acute mountain sickness, high-altitude cerebral edema, or high-altitude pulmonary edema
5. Been on a high-altitude trek 2 weeks prior to this study
6. Has taken acetazolamide 1 week prior to start of trek
7. Has a sulfa allergy
8. Has any type of acute or chronic pulmonary conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Irons, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No ipd to share.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetazolamide Normal Dose | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were enrolled, but no participants were randomized to intervention and no participants received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide Normal Dose | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Edema Before and After Taking Acetazolamide
Description: Edema measured through ultrasound exam
Time Frame: 1 month
Population: No participants were randomized and no participants received intervention.
Arm/Group | Acetazolamide Normal Dose | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Completion of Ultrasound Exams
Description: Time it takes to complete ultrasound exams
Time Frame: 1 month
Population: Participants enrolled but not randomized and did not receive study drug.
Arm/Group | Acetazolamide Normal Dose | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Due to investigator illness, no participants were randomized and no study drug was administered.
Description: Due to investigator illness, no participants were randomized and no study drug was administered.
Arm/Group | Acetazolamide Normal Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to Investigator illness, although participants were enrolled, no participants were randomized to receive interventions and did not receive study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03490916/Prot_SAP_000.pdf